CLINICAL TRIAL: NCT05335226
Title: The Efficacy and Safety of Combined Haploidentical and Umbilical Cord Blood Allogeneic Stem Cell Transplantation in Patients With Acute Leukemia.
Brief Title: Combined Haploidentical and Umbilical Cord Blood Allogeneic Stem Cell Transplantation in Patients With Acute Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220410
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Acute Leukemia
Keywords: Acute Leukemia; haplo-hematopoietic stem cell transplantation (haplo-HSCT); umbilical cord blood stem cell transplantation (UCBT)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haplo-HSCT group (Experimental): 58 patients will be involved in this group
  Interventions: Procedure: haploidentical hematopoietic stem cell transplantation
- Combined haploidentical and umbilical cord blood allogeneic stem cell transplantation group (Experimental): 58 patients will be involved in this group
  Interventions: Procedure: Combined haploidentical and umbilical cord blood allogeneic stem cell transplantation

INTERVENTIONS:
Procedure: Combined haploidentical and umbilical cord blood allogeneic stem cell transplantation — Patients will receive umbilical cord blood allogeneic stem cell transplantation at the same day as the haploidentical stem cell transplantation. (HLA 6-10/10, TNC≥1-3×10-7/Kg)
  Arms: Combined haploidentical and umbilical cord blood allogeneic stem cell transplantation group
Procedure: haploidentical hematopoietic stem cell transplantation — Receive haploidentical hematopoietic stem cell transplantation (HLA 6-10/10)
  Arms: Haplo-HSCT group

SUMMARY:
Allogeneic stem cell transplantation (Allo-HSCT) is the effective and even the only treatment option for acute leukemia. The haplo-hematopoietic stem cell transplantation(haplo-HSCT) and "GIAC" protocol have crossed HLA barrier and helped more patients find donors. However, the engraftment failure and incidence of graft-versus-host disease(GVHD) limit the prognosis of patients who receive the haplo-HSCT. It is believed that Combined haploidentical and umbilical cord blood allogeneic stem cell transplantation improved hematopoietic reconstitution and reduced the incidence of GVHD, there is still no consensus about the efficacy and safety of this kind of therapy. This prospective, randomized and controlled study is to investigate the efficacy and safety of Combined haploidentical and umbilical cord blood allogeneic stem cell transplantation

DETAILED DESCRIPTION:
This prospective, randomized and controlled study is to investigate the efficacy and safety of Combined haploidentical and umbilical cord blood allogeneic stem cell transplantation. Investigators will recruit 116 patients with acute leukemia, with 58 of them entering the haplo-HSCT group and receiving haploidentical hematopoietic stem cell transplantation, while the other 58 entering the combined haploidentical and umbilical cord blood allogeneic stem cell transplantation group and receiving haploidentical and umbilical cord blood allogeneic stem cell transplantation at the same day. Then primary outcomes including overall survival and disease free survival, as well secondary outcomes such as cumulative relapse incidence and cumulative incidence of engraftment will be measured during 12 months after the intervention being finished.

ELIGIBILITY:
Inclusion Criteria:

* Ages 16-65 years inclusive.
* Diagnosed as acute leukemia, planning to receive haplo-HSCT
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2
* Presence of an available haploidentical donor
* Signing written informed consent and agreeing with taking designated umbilical cord blood

Exclusion Criteria:

* Uncontrolled infections less than 4 weeks prior to enrollment
* Secondary malignancy
* Psychiatric illness that would limit compliance with study requirements
* Impairment of heart, hepatic or renal function to such an extent that the patient, in the opinion of the investigator, will be exposed to an excessive risk if entered into this clinical study
* Allergic to blood products
* Other causes which are not suitable for the trial in investigator's consideration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 12 months
  Defined as the survival duration starting at the day of transplantation, terminating at the day of death or the end of follow-up
Disease free survival | 12 months
  Defined as the time starting at the day of transplantation, terminating at the day when the sign of AL is found or the end of follow-up

SECONDARY OUTCOMES:
Cumulative relapse incidence | 12 months
  Defined as the cumulative incidence of relapse after the day of transplantation
Cumulative incidence of engraftment | 12 months
  Neutrophil recovery was defined as an absolute neutrophil count(ANC) of 0.5×10^9/L or more for three consecutive days , while platelet recovery difined as 20×10^9/L or more for seven consecutive days without transfusion
cumulative incidence of acute graft-versus-host disease(GVHD) | 12 months
  Acute graft versus host disease will be diagnosed and graded by modified Glucksberg criteria
cumulative incidence of chronic GVHD at one year | 12 months
  chronic graft versus host disease will be diagnosed and graded by National Institute of Health Consensus (NIH Consensus)
Cumulative Incidence of Infectious Complications | 12 months
  Defined as cumulative incidence of viral, fungal and bacterial infections
Cumulative Incidence of hemorrhagic cystitis | 12 months
  Defined as the cumulative incidence of hemorrhagic cystitis after the day of transplantation
Cumulative Incidence of lymphoproliferative disease | 12 months
  Defined as the cumulative incidence of lymphoproliferative disease after the day of transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Erlie Jiang, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China